CLINICAL TRIAL: NCT02955082
Title: The BARCODE 2 Study - The Use of Genetic Profiling to Guide Prostate Cancer Treatment
Acronym: BARCODE2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); European Research Council (Other); Imperial College Healthcare NHS Trust (Other); Dartford and Gravesham NHS Foundation Trust (Unknown); Maidstone & Tunbridge Wells NHS Trust (Other); East and North Hertfordshire NHS Trust (Other Government); Royal Free Hampstead NHS Trust (Other); Buckinghamshire Healthcare NHS Trust (Other); Barts & The London NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); Yeovil District Hospital NHS Foundation Trust (Other); Northampton General Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4520
Record Dates: First submitted 2016-10-10; First posted 2016-11-04 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hormone Refractory Prostate Cancer
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carboplatin (Experimental): Patients with a germline DNA repair gene mutation identified in part 1 of the study, or who are already known to have a germline mutation will undergo assessment for inclusion in part 2 of the study to receive Carboplatin treatment.
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Intravenous carboplatin infusion every 3 weeks.
  Other Names: Paraplatin

SUMMARY:
Prostate cancer (PrCa) is one of the commonest cancer in men in the Western world. In the United Kingdom (UK), there were over 52,000 new cases diagnosed in 2016-2018 and a lifetime risk of 1 in 8. Research studies have identified several genetic changes that are thought to increase the risk of developing prostate cancer. Some of these genetic changes occur in deoxyribonucleic acid (DNA) repair genes. The BARCODE 2 trial is formed of two parts that aim to investigate how having genetic changes in DNA repair genes can affect response to carboplatin treatment in patients with metastatic castration resistant prostate cancer (mCRPC). In part 1 of the study, the investigators will invite men with mCRPC who have not had genetic testing before to join the study by initially undergoing genetic screening within the study. The DNA repair gene mutation carrier status of enrolled patients will be assessed using a gene panel. If a pathogenic mutation is confirmed in one of these genes, patients will be given the option to proceed to part 2 of the study. In part 2 of the study, men with mCRPC who are known to be carriers of a mutation in DNA repair gene(s) will be assessed for eligibility for treatment on the study with carboplatin chemotherapy. The aim of the study will be to determine how patients with mCRPC and a germline mutation in a DNA repair gene(s) respond to platinum chemotherapy. This study will help researchers to investigate platinum sensitivity of prostate tumours that have developed due to a germline mutation in a DNA repair gene. This study will provide data to use in a larger clinical trial of platinum chemotherapy based on patients' germline genetic signature and/or tumour genetic profile.

DETAILED DESCRIPTION:
Purpose and Design

BARCODE 2 is a single arm, single site phase II trial with the aim to determine the response rate to two cycles of platinum chemotherapy in patients with mCRPC and a germline mutation in a DNA repair gene. Response will be measured with prostate specific antigen (PSA) levels and radiological assessment. The study will be divided into two parts. In part 1 of the study, the DNA repair gene mutation carrier status of enrolled patients will be assessed using a gene panel. Men who are found to carry a pathogenic mutation or are already known to carry a germline mutation can enrol in part 2 of the study and be offered treatment with carboplatin.

Eligibility and Recruitment

Patients with mCRPC which has progressed after docetaxel chemotherapy and androgen receptor-directed therapy (e.g., abiraterone or enzalutamide) may be assessed for eligibility for study entry. Patients who have completed treatment with or are currently undergoing cabazitaxel chemotherapy are also eligible.

Inclusion Criteria

All study participants will be assessed according to the part 1 and/ or part 2 inclusion criteria depending on which part of the study they enter initially (see inclusion/exclusion criteria further below).

Informed Consent

Participants will be given the latest ethically approved BARCODE 2 participant information sheet (PIS) for their consideration. Patients will only be asked to consent to the study after they have had sufficient time to consider the trial, and the opportunity to ask any further questions. Patients who have not had previous genetic testing will sign the part 1 consent form to undergo genetic profiling for a germline mutation in a DNA repair gene. Patients who are found to have a pathogenic mutation in part 1 or who are already known to carry a germline mutation must sign the part 2 consent form prior to undergoing part 2 study related procedures.

Patient Confidentiality

Patients will be asked to consent to their full name being collected at trial entry in addition to their date of birth, hospital number, postcode and National Health Service (NHS) number or equivalent to allow linkage with routinely collected NHS data and ensure accuracy in handling biological samples.

Investigators will ensure that all participants' personal identifier information is kept on a separate log.

Investigators will retain trial documents in strict confidence. Investigators will maintain the confidentiality of participants at all times and will not reproduce or disclose any information to third parties by which participants could be identified (without consent).

Data Protection

The study will comply with all applicable data protection laws.

Subject Withdrawal

Participants may discontinue from the trial at any time at their own request, or they may be discontinued from trial treatment at the discretion of the Principal Investigator (PI). Reasons for discontinuation will include:

* Clinical or radiological disease progression.
* Unacceptable toxicity (e.g. unresolving grade ≥2 neuropathy or neutropenia)
* Any other reason deemed appropriate by investigator. Increases in PSA will not be a criterion for treatment discontinuation in the absence of clinical or radiological progression. Participants who discontinue treatment should continue to be followed up until death.

Post-treatment Follow-up

Follow up data will be collected on all patients entering part 2 of the study who received carboplatin treatment on this trial until death, including cause of death. Survival data will be collected on all participants on the BARCODE 2 trial. Participants who discontinue treatment should continue to be followed up until death.

Discontinuation from Follow-up

If a patient withdraws from further follow-up, a trial deviation form should be submitted to Oncogenetics Team stating whether the patient has withdrawn consent for information to be sent to the Oncogenetics Team or whether they simply no longer wish to attend trial follow up visits. In the very rare event that a patient requests that their data is removed from the study entirely, the implications of this should be discussed with the patient first to ensure that this is their intent and, if confirmed, the Oncogenetics Team should be notified in writing. If this request is received after results have been published the course of action will be agreed between the Sponsor and Independent Data Monitoring and Steering Committee.

Trial Management

A Trial Management Group (TMG) will be set up and will include the Chief Investigator, the Trial Statistician and Trial Manager. Key study personnel will be invited to join the TMG as appropriate to ensure representation from a range of professional groups, including a PI from a Participant Identification Centre (PIC). Membership will include a lay/consumer representative who will receive support and training as deemed necessary. The TMG will meet at regular intervals, and at least annually. The TMG have operational responsibility for the conduct of the trial.

Independent Data Monitoring and Steering Committee (IDMSC)

A joint Independent Data Monitoring and Steering Committee (IDMSC) will be set up to oversee the safety of the trial participants, monitor the data produced by the trial, put these data into overall context and supervise the progress of the trial towards its interim and overall objectives.

Publication and Data Sharing Policy

The main trial results will be published in a peer-reviewed journal, on behalf of all collaborators. Anonymised data can be applied for via the Data Access Committee.

ELIGIBILITY:
Inclusion Criteria:

All study participants will be assessed according to the part 1 and/ or part 2 inclusion criteria depending on which part of the study they enter initially.

For Part 1 (genetic screening) of the study:

1. Age ≥ 18 years.
2. Recorded diagnosis of prostate cancer with or without histological confirmation. Patients who have not previously undergone a prostate (or metastatic) biopsy but are confirmed to have a raised PSA (>80ng/ml at any time), metastatic disease on imaging and have undergone treatment for mCRPC are eligible.
3. Castration-resistant disease defined as biochemical or radiological progression on/after treatment with orchidectomy or LHRH analogues as per PCWG3 criteria.
4. Confirmed metastatic disease on conventional imaging methods such as CT, bone scan or PET imaging.
5. Current or previous treatment includes at least one of the following:

   1. Docetaxel (either in hormone sensitive or resistant setting; Patients who have completed treatment with or are currently undergoing Cabazitaxel chemotherapy are also eligible)
   2. Androgen receptor-directed therapy (e.g., Enzalutamide, Abiraterone)
6. Adequate renal function measured by calculated GFR (Cockcroft-Gault) >30ml/min. If a participant had renal dysfunction that is expected to improve, they may be considered for part 1 of the study.
7. Adequate haematological function to allow study entry in line with local hospital practice or at the investigator's discretion.
8. WHO performance status 0-2 as assessed and documented by study doctor.
9. Life expectancy >12 weeks
10. Participants with stable, treated brain metastases will be eligible providing informed consent can be given and that other sites of measurable disease are present
11. The subject is capable of understanding and complying with the protocol requirements and has signed the BARCODE 2 informed consent form.

In addition to the above, for Part 2 of the study:

1. Confirmed pathogenic germline mutation in a DNA repair gene. (Participants with a known germline mutation will need to provide a report from the external laboratory where genetic testing was carried out)
2. Previous treatment with docetaxel and androgen receptor-directed therapy (e.g., abiraterone or enzalutamide) with documented disease progression prior to entry to part 2 (rising PSA and/or radiographic progression). Patients previously treated with cabazitaxel and who have documented disease progression are also eligible.
3. Adequate haematological function: Haemoglobin (Hb) ≥8.0g/dL, neutrophil count ≥1.5x109/L and platelets ≥100x109/L.
4. Adequate liver function: Total bilirubin ≤1.5 x upper limit of normal (ULN) except for participants with known Gilbert's syndrome; AST and ALT ≤ 2.5x ULN in the presence of liver metastases.
5. Adequate renal function: creatinine clearance >30ml/min measured by a glomerular filtration rate (GFR) clearance test. If a measured GFR test is not available, then calculated GFR is acceptable (measured GFR must be carried out by cycle 2 of carboplatin).

Exclusion Criteria (for part 1 and 2):

1. Critical organ metastases (e.g. spinal metastases with risk of cord compression) as documented on most recent imaging report.
2. Participants with bleeding tumours.
3. Previous treatment with a platinum chemotherapy drug for prostate cancer.
4. Previous treatment with a PARP inhibitor
5. Participants with a history of severe allergic reaction to carboplatin or other platinum-containing compounds
6. Exposure to yellow fever vaccine in the previous 6 months.
7. Participants unfit for chemotherapy or those with ongoing neuropathy >grade 1 (sensory or motor) according to NCI CTCAE V4.02.
8. Known and documented hearing impairment
9. Other active malignancies or previous malignancies likely, in the PI's opinion, to impact on management of mCRPC.
10. Significant documented cardiovascular disease: severe/unstable angina, myocardial infarction less than 6 months prior to trial entry, arterial thrombotic events less than 6 months prior to trial entry, clinically significant cardiac failure requiring treatment (NYHA II-IV).
11. Cerebrovascular disease (CVA or TIA) in the preceding 2 years to entry to Part 2 of study.
12. Presence of symptomatic brain metastases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must be male at birth.
Enrollment: 305 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic Treatment Response | 6 weeks
  Response rate to two cycles of platinum chemotherapy in patients with mCRPC and germline DNA repair gene mutations using the modified response evaluation criteria in solid tumours (RECIST) 1.1 criteria. In participants with bone only metastatic disease, response will be recorded as having 'new lesions' or 'no new lesions' (as per the Prostate Cancer Working Group 3 (PCWG3) guidance). Participants with no new bone lesions will be deemed as having stable disease. These participants can respond by PSA as defined below.
Radiographic Treatment Response | 9 weeks
  Response rate to three cycles of platinum chemotherapy in patients with mCRPC and germline DNA repair gene mutations via bone scan assessment. In participants with bone only metastatic disease, response will be recorded as having 'new lesions' or 'no new lesions' (as per PCWG3 guidance). Participants with no new bone lesions will be deemed as having stable disease. These participants can respond by PSA as defined below.
Biochemical Treatment Response | 6 weeks
  Reduction of more than 50% in PSA levels in response to two cycles of platinum chemotherapy in patients with mCRPC and germline DNA repair gene mutations.

SECONDARY OUTCOMES:
Overall survival of men with mCRPC and germline DNA repair gene mutations | This will be evaluated 3 months after end of study treatment
  Overall survival of patients with mCRPC and a DNA repair gene mutation treated with carboplatin.
Progression-free survival of men with mCRPC and germline DNA repair gene mutations | This will be evaluated 3 months after end of study treatment
  Progression free survival of patients with mCRPC and a DNA repair gene mutation treated with carboplatin.
Incidence of germline DNA repair gene mutations in a population of mCRPC cases | Through study completion, up to 3 years
  Incidence of germline DNA repair gene mutations will be calculated from the rate of pathogenic mutations observed in the group of men who undergo genetic profiling within part 1 of the study.
Bone scan response | Through study completion, up to 3 years
  Bone scan response (new lesion vs. no new lesions) at each time point in patients with bone-only metastatic disease.
Cause specific survival | This will be evaluated 3 months after end of study treatment
  Cause specific survival from date of first diagnosis of prostate cancer in patients with DNA repair gene mutations.
Radiographic progression free survival | This will be evaluated 3 months after end of study treatment
  Radiographic Progression free survival will be measured from the date of trial entry to the first occurrence of radiographic progression or death.
Time to radiographic progression | This will be evaluated 3 months after end of study treatment
  Time to radiographic progression will be measured from the date of trial entry to the first occurrence of radiographic progression.
PSA objective responses | This will be evaluated 3 months after end of study treatment
  PSA response and PSA progression are defined according to the consensus guidelines of the Prostate Cancer Working Group 3 (PCWG3).

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, FRCP, FRFR, Principal Investigator — Institute of Cancer Research and Royal Marsden Hospital
Locations (1):
- Institute of Cancer Research and Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Data Access Committee.

REFERENCES:
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579